CLINICAL TRIAL: NCT03366753
Title: Impact of Intravascular Fluid Resuscitation for Acute Normovolemic Hemodilution on Blood Viscosity and Oxygen Delivery in Coronary Artery Bypass Graft Surgery
Brief Title: Impact of Acute Normovolemic Hemodilution on Blood Viscosity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: KUH1160102
Record Dates: First submitted 2017-11-28; First posted 2017-12-08 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Ischemic Heart Disease; Coronary Artery Disease
Keywords: acute normovolemic hemodilution; coronary artery bypass graft surgery; hydroxyethyl starch; blood viscosity
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Acute normovolemic hemodilution consists of phlebotomy and intravascular volume resuscitation by using crystalloid/colloid in a same amount of phlebotomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute normovolemic hemodilution (Experimental): acute normovolemic hemodilution by using hydroxyethyl starch
  Interventions: Procedure: acute normovolemic hemodilution; Procedure: In-vitro hemodilution
- In-vitro hemodilution (Experimental): adding additional hydroxyethyl starch for achieving further 30% dilution of whole blood sample which already underwent ANH of 4-6 ml/kg.
  Interventions: Procedure: In-vitro hemodilution

INTERVENTIONS:
Procedure: acute normovolemic hemodilution — acute normovolemic hemodilution (ANH) is performed by using 5 ml/kg of blood salvage and intravenously administering 5 ml/kg of balanced hydroxyethystarch 130/0.42 (Tetraspan™) for 15 min
  Arms: Acute normovolemic hemodilution
Procedure: In-vitro hemodilution — Blood sample after ANH 5 ml/kg undergoes further 30% in-vitro dilution by adding 1-1.5 ml hydroxyethystarch 130/0.42

SUMMARY:
Acute normovolemic hemodilution (ANH) has long been employed for reducing allogenic blood transfusion for cardiac surgery, and hydroxyethyl starch has been used as an intravenous replacement fluid during ANH procedure. However, possible impact of ANH employing HES on blood viscosity and oxygen delivery have not been well investigated in patients undergoing off-pump coronary artery bypass (OPCAB) surgery .

Anesthesia is induced and maintained by using propofol-remifentanil-rocuronium in OPCAB surgery (n=21). ANH is performed by using 5 ml/kg of blood salvage and administering 5 ml/kg of balanced HES 130/0.42 (Tetraspan™) for 15 min during vascular graft harvesting. For the present study, three arterial blood samples (3 ml each) are taken before (Sample 1) and after ANH (sample 2 and 3) and they are stored in 3 tubes. Sample 3 (in tube) undergoes further 30% in-vitro dilution by adding 1-1.5 ml HES. By using a scanning capillary tube viscometer (Hemovister™), Blood viscosity at low shear rate (5/sec) of the three samples are determined. By using a formula with blood viscosity and hematocrit, tissue O2 delivery index (TODI, = hematocrit/viscosity at 5/sec) is calculated.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing off-pump coronary artery bypass graft surgery

Exclusion Criteria:

* Preoperative anemia
* LV ejection fraction < 50%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
blood viscosity at shear rate 5/sec | 5 min after acute normovoelmic hemodilution, 5 min after in-vitro dilution
  By using a scanning capillary tube viscometer (Hemovister™), Blood viscosity at shear rate 5/sec of the three samples are determined
hematocrit/blood viscosity at 5/sec | 5 min after acute normovoelmic hemodilution, 5 min after in-vitro dilution
  oxygen delivery index calculated with a formula (= hematocrit/blood viscosity)

SECONDARY OUTCOMES:
blood viscosity at shear rate 300/sec | 5 min after acute normovoelmic hemodilution, 5 min after in-vitro dilution
  By using a scanning capillary tube viscometer (Hemovister™), Blood viscosity at shear rate 300/sec of the three samples are determined
Hematocrit/viscosity at shear rate 300/sec | 5 min after acute normovoelmic hemodilution, 5 min after in-vitro dilution
  oxygen delivery index calculated with a formula (= hematocrit/blood viscosity)
Coagulation profiles in ROTEM | 5 min after acute normovoelmic hemodilution, 5 min after in-vitro dilution
  clot formation time in extem, MCF in extemA5 in fibtem,

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD PhD, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No